CLINICAL TRIAL: NCT02063672
Title: A Prospective, Multicenter, Single-Blind, Randomized, Controlled Trial Comparing the Lutonix® Drug Coated Balloon vs. Standard Balloon Angioplasty for Treatment of Femoropopliteal In-Stent Restenosis
Brief Title: Lutonix® Drug Coated Balloon vs. Standard Balloon Angioplasty for Treatment of Femoropopliteal In-Stent Restenosis
Acronym: SFA ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL0018-01
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Femoral Artery Stenosis; Femoral Artery Occlusion; Restenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutonix DCB (Experimental): Lutonix Paclitaxel Drug Coated Balloon
  Interventions: Device: Lutonix DCB
- PTA Catheter (Active Comparator): Standard Uncoated Balloon Angioplasty Catheter
  Interventions: Device: Standard Uncoated Balloon Angioplasty Catheter

INTERVENTIONS:
Device: Lutonix DCB
  Arms: Lutonix DCB
Device: Standard Uncoated Balloon Angioplasty Catheter — PTA Catheter
  Arms: PTA Catheter

SUMMARY:
To assess the safety and efficacy of the Lutonix Drug Coated Balloon for treatment of femoropopliteal artery (SFA) in-stent restenosis (ISR).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or non-pregnant female ≥18 years of age
2. Rutherford Clinical Category 2-4
3. Significant (≥ 50%) restenosis of a previous bare (not covered and not drug-eluting) nitinol stent(s) in the femoropopliteal artery
4. Lesion measures between 4 and 18 cm
5. Target vessel diameter between ≥4 and ≤6 mm and able to be treated with available device size matrix
6. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography
7. Successful crossing and predilatation of the target lesion with a guidewire
8. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography that has not previously been (nor planned to be) revascularized
9. No other prior vascular or surgical interventions within 2 weeks before and/or planned 30 days after the protocol treatment

Key Exclusion Criteria:

1. Life expectancy of <1 year
2. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study NOTE: Enrollment in another drug or device clinical trial during the follow up period is not allowed
3. History of stroke within 3 months
4. History of MI, thrombolysis or angina within 2 weeks of enrollment
5. Prior vascular surgery of the index limb, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion
6. Target lesion involves a previously placed covered stent or drug-eluting stent
7. Grade 4 or 5 stent fracture (mal-aligned components or trans-axial spiral configuration) in the restenotic stent
8. Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication
9. Known inadequate distal outflow (>50 % stenosis of distal popliteal and/or all three tibial vessels), or planned future treatment of vascular disease distal to the target lesion
10. Intended use of adjunctive treatment modalities (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, stents, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-03; Primary Completion 2017-02-13 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena, MD, Principal Investigator — Yale University
Locations (20):
- United States (20):
  - Cardiology Associates, Fairhope, Alabama
  - Yale University, New Haven, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Radiology and Imaging Specialists of Lakeland, P.A., Lakeland, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - Northwestern University, Evanston, Illinois
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - Metropolitan Hospital d/b/a Metro Health Hospital, Wyoming, Michigan
  - Minneapolis Radiology and Vascular Research Foundation, Plymouth, Minnesota
  - Hattiesburg Clinic, PA, Hattiesburg, Mississippi
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - Kansas City Vascular Foundation, North Kansas City, Missouri
  - Hunterdon Cardiovascular Associates, Flemington, New Jersey
  - Rex Hospital, Inc., Raleigh, North Carolina
  - TriHealth, Inc., Cincinnati, Ohio
  - The Miriam Hospital - A Lifespan Partner, Providence, Rhode Island
  - Wellmont Cardiology Services, Inc., Kingsport, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lutonix DCB: Lutonix Paclitaxel Drug Coated Balloon
  Lutonix DCB
Period: Overall Study
Arm/Group | Lutonix DCB | PTA Catheter
Started | 53 | 29
Completed | 18 | 7
Not Completed | 35 | 22
Not completed — Ongoing Follow-up | 27 | 14
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix DCB | PTA Catheter | Total
Number analyzed (Participants) | 53 | 29 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.35) | 67.0 (8.64) | 68.2 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 30 | 12 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 45 | 23 | 68
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Primary Patency at 1 Year
Description: Primary patency is defined as freedom from clinically driven target lesion restenosis (TLR) and from Binary Restenosis.
Time Frame: 12 Months
Population: All subjects who completed a 12-Month follow-up visit
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 49 | 23
Percentage of Participants | 67.0 [50.5 to 79.1] | 49.5 [26.2 to 69.2]

2. Primary Outcome: Percentage of Participants Without Primary Safety Events
Description: Primary Safety Events include: All Cause Perioperative (≤30 day) Death, Index Limb Amputation, Index Limb Reintervention and Index Limb Related Death at 1 Year
Time Frame: 12 Months
Population: All participants with 12-month evaluable data for the primary safety endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 40 | 16
Percentage of Participants | 72.8 [58.4 to 82.9] | 64.0 [42.0 to 79.5]

3. Secondary Outcome: Percentage of Participants With Device Success
Description: Device success is defined as, on a per device basis, the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the study system.
Time Frame: During the Index Procedure (90 mins)
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 53 | 28
Percentage of Participants | 98.1 [89.9 to 100.0] | 100 [87.7 to 100.0]

4. Secondary Outcome: Percentage of Participants With Technical Success
Description: Technical success of the balloon procedure is defined as the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion and a successful withdrawal of the study system with the achievement of < 30% residual percent stenosis without deployment of a bail-out stent.
Time Frame: During the Index Procedure (90 mins)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 27
Percentage of Participants | 66.0 [51.2 to 78.8] | 77.8 [57.7 to 91.4]

5. Secondary Outcome: Percentage of Participants With Procedural Success
Description: Procedural Success is defined as attainment of ≤30% residual stenosis in the treatment area by independent core lab analysis without major adverse events (defined as occurrence of death, amputation of the target limb, or repeat revascularization of the target lesion) during the index procedure and through the hospital stay.
Time Frame: During the Index Procedure (90 mins)
Population: All participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 27
Percentage of Participants | 70.0 [55.4 to 82.1] | 77.8 [57.7 to 91.4]

6. Secondary Outcome: Percentage of Participants With Primary Patency at 6 and 12 Months
Description: Primary Patency is defined as Freedom from CEC-adjudicated Clinically-Driven TLR and from Core laboratory-adjudicated Binary Restenosis. Binary restenosis is based on threshold Doppler peak systolic velocity ratio (PSVR) ≥ 2.5 (together with waveform analysis & color mosaic appearance) or based on angiographic ≥ 50% diameter stenosis (if angiography is performed although not required per protocol).
Time Frame: 6 months and 12 months
Population: All participants with evaluable data at each time point.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 43 | 20
Percentage of Participants
  6 Months | 92.1 [80.2 to 96.9] | 77.0 [53.1 to 89.8]
  12 Months: number analyzed (Participants) | 32 | 8
  12 Months | 67.0 [50.5 to 79.1] | 37.1 [16.1 to 58.4]

7. Secondary Outcome: Percentage of Participants With Secondary Patency at 6 Months and 12 Months
Description: Secondary patency is defined as the absence of Binary Restenosis as adjudicated by the blinded, independent core laboratory, independent of whether or not patency is re-established via an endovascular procedure.
Time Frame: 6 months and 12 months
Population: All participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 33 | 10
Percentage of Participants
  6 Months | 90.9 [75.7 to 98.1] | 60.0 [26.2 to 87.8]
  12 Months: number analyzed (Participants) | 31 | 10
  12 Months | 74.2 [55.4 to 88.1] | 80.0 [44.4 to 97.5]

8. Secondary Outcome: Percentage of Participants Without Clinically Driven Target Lesion Revascularization (TLR)
Description: Clinically-driven TLR is defined as revascularization of the target vessel with evidence of target vessel diameter stenosis >50% determined by duplex ultrasound or angiography and new distal ischemic signs (worsening ABI or worsening Rutherford Category associated with the target limb or due to clinical symptoms), OR revascularization of a target vessel with an in-lesion diameter stenosis of >70% by angiography, in the absence of the previously mentioned ischemic signs or symptoms.
Time Frame: 6 months and 12 months
Population: All participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 26
Percentage of Participants
  6 Months | 94.3 [83.4 to 98.1] | 96.4 [77.2 to 99.5]
  12 Months: number analyzed (Participants) | 43 | 16
  12 Months | 78.6 [64.7 to 87.5] | 64.0 [42.0 to 79.5]

9. Secondary Outcome: Percentage of Participants Without Target Lesion Revascularization (TLR)
Description: TLR is defined as any repeat revascularization procedure (percutaneous or surgical) of the original target lesion site.
Time Frame: 6 months and 12 months
Population: All participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 26
Percentage of Participants
  6 Months | 94.3 [83.4 to 98.1] | 92.7 [73.9 to 98.1]
  12 Months: number analyzed (Participants) | 43 | 16
  12 Months | 78.6 [64.7 to 87.5] | 64.0 [42.0 to 79.5]

10. Secondary Outcome: Percentage of Participants With Sustained Clinical Benefit Compared to Baseline
Description: Sustained clinical benefit is defined as an improvement in Rutherford Classification compared to baseline and freedom from target vessel revascularization. The Rutherford classification is a clinical means of describing peripheral artery disease along a seven-stage scale, with stage 0 representing asymptomatic presentation and stage 6 representing severe ischemic ulcers or frank gangrene. A decrease in units on the scale represents improvement in clinical symptoms.
Time Frame: 6 months and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 49 | 22
Percentage of Participants
  6 Months | 69.4 [54.6 to 81.7] | 59.1 [36.4 to 79.3]
  12 Months | 61.2 [46.2 to 74.8] | 50.0 [28.2 to 71.8]

11. Secondary Outcome: Change of Rutherford Classification From Baseline
Description: The Rutherford classification is a clinical means of describing peripheral artery disease along a seven-stage scale, with stage 0 representing asymptomatic presentation and stage 6 representing severe ischemic ulcers or frank gangrene. A decrease in units on the scale represents improvement in clinical symptoms.
Time Frame: 6 months and 12 months
Population: All patients with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 49 | 22
units on a scale
  6 Months | -1.7 (1.26) | -1.5 (1.41)
  12 Months | -1.6 (1.17) | -1.9 (1.06)

12. Secondary Outcome: Change of Resting Ankle Brachial Index (ABI) From Baseline
Description: The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium).
Time Frame: 6 months and 12 months
Population: All participants with evaluable data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 39 | 17
ratio
  6 Months: number analyzed (Participants) | 39 | 15
  6 Months | 0.20 (0.20) | 0.25 (0.30)
  12 Months: number analyzed (Participants) | 38 | 17
  12 Months | 0.16 (0.20) | 0.16 (0.24)

13. Secondary Outcome: Change in Walking Impairment Questionnaire From Baseline
Description: The Walking Impairment Questionnaire (WIQ) is a validated questionnaire that evaluates walking ability with a focus on walking distance, walking speed, and the ability to climb stairs. Participants answer each item on a Likert scale from 0 for "unable to do" to 4 for "no difficulty", and each response is weighted based on the difficulty of the task. The overall score is determined by dividing the weighted answers by the maximum possible weighted score and multiplying by 100. The overall score ranges from 0-100 with lower scores indicating lower performance.
Time Frame: 6 months and 12 months
Population: All participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 49 | 23
units on a scale
  6 Months: number analyzed (Participants) | 49 | 22
  6 Months | 14.9 (28.6) | 16.0 (38.3)
  12 Months | 12.7 (22.6) | 12.7 (27.7)

14. Secondary Outcome: Change in Quality of Life From Baseline
Description: EQ-5D is a standardized tool to assess patient-reported mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, or slight, moderate, severe, or extreme problems. Patients choose the appropriate level in each of the 5 dimensions, which results in a 1-digit number for each dimension. The digits for the 5 dimensions are converted into a single EQ-5D™ index score based on a set of population-based preference weights. For the U.S. general population, possible EQ-5D™ index scores range from -0.11 (i.e., 33333) to 1.0 (i.e., 11111) on a scale where 0.0 = death and 1.0 = perfect health. A downloadable scoring file is available at: https://www.ahrq.gov/rice/EQ5Dscore.htm.
  The EQ VAS records a patient's self-rated health on a vertical visual analogue scale, where the endpoints are labeled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). A higher VAS value indicates a higher quality of life.
Time Frame: 6 months and 12 Months
Population: All participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 49 | 23
units on a scale
  6 Months - EQ5D Index: number analyzed (Participants) | 47 | 22
  6 Months - EQ5D Index | 0.1 (0.18) | 0.0 (0.24)
  12 Months - EQ5D Index | 0.0 (0.19) | 0.0 (0.23)
  6 Months - EQ5D VAS: number analyzed (Participants) | 47 | 22
  6 Months - EQ5D VAS | -2.0 (23.1) | 0.3 (23.2)
  12 Months - EQ5D VAS: number analyzed (Participants) | 48 | 23
  12 Months - EQ5D VAS | 2.9 (23.0) | 0.5 (24.8)

15. Secondary Outcome: Percentage of Participants Without Major Vascular Complications (≤30 Day)
Description: Freedom from major vascular complications at 30 days follow-up
Time Frame: 30 Days
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 52 | 28
Percentage of Participants | 98.1 [89.7 to 100.0] | 92.9 [76.5 to 99.1]

16. Secondary Outcome: Percentage of Participants Without All-Cause Death
Description: Mortality from any cause.
Time Frame: 1 month, 6 months, and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 52 | 28
Percentage of Participants
  1 Month | 100 [NA to NA] — 100% value, CI not applicable | 100 [NA to NA] — 100% value, CI not applicable
  6 Months: number analyzed (Participants) | 52 | 27
  6 Months | 100 [NA to NA] — 100% value, CI not applicable | 96.4 [77.2 to 99.5]
  12 Months: number analyzed (Participants) | 49 | 23
  12 Months | 100 [NA to NA] — 100% value, CI not applicable | 96.4 [77.2 to 99.5]

17. Secondary Outcome: Percentage of Participants Without Major Limb Amputation
Description: Major limb amputation is defined as amputation of the lower limb above the ankle.
Time Frame: 1 month, 6 months, and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 52 | 28
Percentage of Participants
  1 Month | 100 [NA to NA] — 100% Value, CI not calculable | 100 [NA to NA] — 100% Value, CI not calculable
  6 Months: number analyzed (Participants) | 52 | 27
  6 Months | 100 [NA to NA] — 100% Value, CI is not needed | 100 [NA to NA] — 100% Value, CI is not needed
  12 Months: number analyzed (Participants) | 49 | 23
  12 Months | 100 [NA to NA] — 100% Value, CI not calculable | 100 [NA to NA] — 100% Value, CI not calculable

18. Secondary Outcome: Percentage of Participants Without Minor Limb Amputation
Description: Minor limb amputation is defined as amputation of a part of the foot below the ankle.
Time Frame: 1 month, 6 months, and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 52 | 28
Percentage of Participants
  1 Month | 100 [NA to NA] — 100% Value, CI not calculable | 100 [NA to NA] — 100% Value, CI not calculable
  6 Months: number analyzed (Participants) | 52 | 26
  6 Months | 100 [NA to NA] — 100% Value, CI not calculable | 96.4 [77.2 to 99.5]
  12 Months: number analyzed (Participants) | 49 | 26
  12 Months | 100 [NA to NA] — 100% Value, CI not calculable | 96.4 [77.2 to 99.5]

19. Secondary Outcome: Percentage of Participants Without Target Vessel Revascularizations (TVR)
Description: A TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel.
Time Frame: 1 month, 6 months, and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 28
Percentage of Participants
  1 Month | 96.2 [85.7 to 99.0] | 100 [NA to NA] — 100% Value, CI not calculable
  6 Months: number analyzed (Participants) | 47 | 25
  6 Months | 90.5 [78.6 to 95.9] | 92.7 [73.9 to 98.1]
  12 Months: number analyzed (Participants) | 37 | 14
  12 Months | 76.7 [62.6 to 86.0] | 64.0 [42.0 to 79.5]

20. Secondary Outcome: Percentage of Participants Without Any Target Limb Reinterventions
Description: Any surgical intervention in the target limb.
Time Frame: 1 month, 6 months, and 12 months
Population: All participants with evaluable data
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 50 | 28
Percentage of Participants
  1 Month | 96.2 [85.7 to 99.0] | 100 [NA to NA] — 100% Value, CI not calculable
  6 Month: number analyzed (Participants) | 46 | 25
  6 Month | 88.5 [76.2 to 94.7] | 92.7 [73.9 to 98.1]
  12 Month: number analyzed (Participants) | 35 | 14
  12 Month | 72.8 [58.4 to 82.9] | 64.0 [42.0 to 79.5]

ADVERSE EVENTS:
Time Frame: Up to 36 Months
Arm/Group | Lutonix DCB | PTA Catheter
All-Cause Mortality (participants affected / at risk) | 5/53 | 3/29
Serious Adverse Events (participants affected / at risk) | 44/53 | 17/29
Other Adverse Events (participants affected / at risk) | 21/53 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix DCB (N=53) | PTA Catheter (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Thrombosis in device (General disorders) | 2 (2) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 15 (19) | 8 (12)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
chronicl total occlusion of anterior tibial artery (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 3 (3) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 8 (9) | 6 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 7 (8) | 4 (5)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix DCB (N=53) | PTA Catheter (N=29)
Device occlusion (General disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 6 (9) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Femoral artery dissection (Vascular disorders) | 4 (4) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 4 (4) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT02063672/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02063672/SAP_001.pdf